CLINICAL TRIAL: NCT00141726
Title: Soluble Tumor Necrosis Factor Receptor: Enbrel (Etanercept) for the Treatment of Sub-Acute Pulmonary Dysfunction Following Allogeneic Stem Cell Transplantation. A Phase II Study
Brief Title: Study of Enbrel (Etanercept) for the Treatment Sub-Acute Pulmonary Dysfunction After Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 3-31; IRBMED 2003-0590 and HUM 46747 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Lung Injury, Acute; Respiratory Distress Syndrome, Adult; Bronchiolitis Obliterans
Keywords: Enbrel; Stem Cell Transplantation; Lung Injury
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Bronchiolitis Obliterans; Lung Injury | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- etanercept treatment (Experimental): Etanercept for lung injury
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept will be given on an open label, single arm basis to patients with non-infectious, sub-acute lung injury. 0.4 mg/kg/dose to a maximum of 25 mg, subcutaneously, twice weekly, for a total of 24 dosages.
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to determine the effectiveness of etanercept in the treatment of patients with sub-acute lung injury following a bone marrow transplant. This study will also examine the toxicity of treatment with etanercept as well as whether there is an improved quality of life in these patients.

DETAILED DESCRIPTION:
Lung or breathing problems can develop several months to years following a bone marrow transplant. In some cases, these breathing problems develop without any signs of germs or infection in the lungs. The name for this type of breathing problem is called "Sub-Acute Lung Injury". Sub-acute lung injury often develops many months, even years following a bone marrow transplant. It is often characterized by shortness of breath, cough, wheezing and fatigue.

Sub-acute lung injury can either lead to the formation of scar tissue in the lungs (making it difficult to take deep breaths), or it can cause the lungs to get weak (making people feel out of breath easily). Approximately 25 - 50% of patients with sub-acute lung injury may eventually die from the damage in their lungs. Typically, such patients die from infections that develop inside the damaged lungs.

In this study, treatment with an experimental drug called Etanercept will be used. (Enbrel). The physicians feel there is the possibility that Etanercept may help improve breathing. Breathing ability will be assessed prior to treatment as well as during and after treatment so that comparisons can be made.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic bone marrow, cord blood, or peripheral blood stem cell transplants are eligible
* Age >6 years and able to complete pulmonary function testing
* Patients with evidence of sub-acute, non-infectious pulmonary dysfunction (OLD or RLD)
* Recipients of sub-ablative transplant regimens are eligible
* Recipients of donor leukocyte infusions (DLI) post-transplant are eligible
* Patients must be > 100 days post transplant

Exclusion Criteria:

* Patients with hypotension requiring inotropic agents other than dopamine < 5mcg/ kg/ minute for blood pressure support.
* Patients with a positive quantitative bacterial culture from the BAL fluid (≥ 104 CFU/ ml is considered positive)
* Patients whose BAL fluid is positive for significant bacterial pathogens or pathogenic nonbacterial microorganisms (as defined by protocol) by special stain, culture or PCR analysis
* Patients who are enrolled on a phase I or phase II trial for the prophylaxis or treatment of GVHD (acute or chronic) within 7 days of study entry.
* Patients with known hypersensitivity to etanercept.
* Patients who are pregnant.
* Patients with CMV seropositivity at the time of study entry. Testing may include wither CMV PCR analysis or CMV pp65 testing.
* Evidence for multi-system organ failure.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Yanik, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- The University of Michigan Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Yanik GA, Mineishi S, Levine JE, Kitko CL, White ES, Vander Lugt MT, Harris AC, Braun T, Cooke KR. Soluble tumor necrosis factor receptor: enbrel (etanercept) for subacute pulmonary dysfunction following allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Jul;18(7):1044-54. doi: 10.1016/j.bbmt.2011.11.031. Epub 2011 Dec 10. PMID 22155140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from the Blood and Marrow Stem Cell Program at the University of Michigan Medical Center between 2001 and 2008, all subjects having received an allogeneic Stem Cell Transplant (SCT) at least 100 days before study entry.
Period: Overall Study
Arm/Group | Etanercept Treatment
Started | 34
Completed | 31
Not Completed | 3
Not completed — Completed <50% Scheduled Dosing | 3

BASELINE CHARACTERISTICS:
Population: All patients enrolled that received at least one scheduled dose.
Arm/Group | Etanercept Treatment
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 39 [8 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Diagnosis [Number; unit: participants]
  AML/MDS/MF | 16
  Acute Lymphoblastic Leukemia (ALL) | 3
  Chronic Mylogenous Leukemia (CML) | 5
  NHL/CLL | 6
  Myeloma | 2
  Nonmalignant | 2
Human Leukocyte Antigen (HLA) Match [Number; unit: participants]
  HLA Matched | 31
  Mismatch | 3
Cell Source [Number; unit: participants] — Cell source for transplant.
  participants
    Pluripotent Stem Cell (PSC) | 25
    Marrow | 9
Donor Type [Number; unit: participants]
  Matched Related Donor (MRD) | 22
  Unrelated Donor (URD) | 12
Chronic Graft Versus Host Disease (GVHD) Present [Number; unit: participants]
  Yes | 34
  No | 0
Lung Injury Pattern [Number; unit: participants]
  Restrictive | 9
  Obstructive | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a Greater Than or Equal to 10% Improvement in FEV1, or FVC, and DLCO
Description: Response was defined as a greater than or equal to 10% improvement in the absolute value for FEV1 (for obstructive defects) or FVC (for restrictive defects), and DLCO (Diffusing Capacity of the Lungs for Carbon Monoxide) .
Time Frame: week 12 post therapy
Population: 34 subjects were enrolled. Thirty-one of 34 subjects were evaluable for response, with three subjects completing <50% of scheduled dosing.
Measure: Number; unit: percent evaluable participants
Arm/Group | Etanercept Treatment
Number analyzed (Participants) | 31
percent evaluable participants
  ≥10% Improvement in FEV1 / FVC | 32
  ≥10% Improvement in DLCO | 16

2. Secondary Outcome: Percentage of Participants That Experience Grade 3 to 4 Adverse Events
Description: To evaluate the toxicity of etanercept therapy in patients with sub-acute lung injury > 100 days post transplant, the percent incidence of grade 3 to 4 adverse events among evaluable patients was calculated.
Time Frame: continuously (and week 4, week 8 and week 12, week 20)
Population: 34 subjects were enrolled and evaluated for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept Treatment
Number analyzed (Participants) | 34
percentage of participants
  Incidence of Grad 3 to 4 Infection | 14
  Incidence of Grade 3 to 4 Electrolyte Toxicities | 11
  Incidence of Grade 3 to 4 Hyperglycemia | 8
  Incidence of Grade 3 to 4 Renal/GU Toxicities | 6
  Incidence of Grade 3 to 4 Hepatic Toxicities | 6
  Incidence of Grade 3 to 4 Pain | 6
  Incidence of Grade 3 to 4 Hypertension | 3
  Incidence of Grade 3 to 4 GI Toxicities | 3
  Incidence of Grade 3 to 4 CNS Toxicities | 3
  Incidence of Grade 3 to 4 Thrombocytopenia | 3

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected for each patient from time of administration of the first dose of drug up to 28 days after the final dose of study drug.
Description: Serious Adverse Events (SAEs) are defined as Grade 4 or 5 (Adverse events will use the descriptions and grading scales found in the revised National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 2.0.) non-pulmonary toxicities.
Arm/Group | Etanercept Treatment
Serious Adverse Events (participants affected / at risk) | 5/34
Other Adverse Events (participants affected / at risk) | 21/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept Treatment (N=34)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacteremia/Infection (Infections and infestations) | 1 (1)
AML Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept Treatment (N=34)
Anemia (Blood and lymphatic system disorders) | 7 (7)
anorexia (Metabolism and nutrition disorders) | 2 (2)
blisters (Skin and subcutaneous tissue disorders) | 2 (2)
chills (General disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2)
bronchoalveolar lavage - positive for bacteria (Respiratory, thoracic and mediastinal disorders) | 4 (6)
cushingoid appearance (Endocrine disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (3)
dizzyness (Nervous system disorders) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
DVT (Vascular disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
dysuria (Renal and urinary disorders) | 2 (2)
Ecchymosis (Vascular disorders) | 2 (2)
elevated Alkaline Phoshpatase (Investigations) | 8 (8)
elevated ALT (Investigations) | 12 (12)
elevated AST (Investigations) | 12 (12)
elevated Creatinine (Investigations) | 8 (8)
elevated T-bili (Investigations) | 3 (3)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fatigue (General disorders) | 4 (4)
fever (General disorders) | 2 (2)
gastroenteritis (Gastrointestinal disorders) | 2 (2)
headache (Nervous system disorders) | 2 (2)
hematuria (Renal and urinary disorders) | 3 (4)
hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 16 (16)
hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
hyperphosphatemia (Metabolism and nutrition disorders) | 4 (4)
hypertension (Vascular disorders) | 4 (5)
hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
hypoalbuminemia (Metabolism and nutrition disorders) | 8 (8)
hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
hypokalemia (Metabolism and nutrition disorders) | 4 (4)
hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
hyponatremia (Metabolism and nutrition disorders) | 4 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
hypotension (Vascular disorders) | 2 (2)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
insomnia (Psychiatric disorders) | 3 (3)
irregular heart beat (Cardiac disorders) | 2 (2)
pruitis (Skin and subcutaneous tissue disorders) | 4 (4)
leg edema (General disorders) | 4 (4)
leukopenia (Blood and lymphatic system disorders) | 3 (3)
lower extremity soreness (General disorders) | 2 (2)
lymphopenia (Blood and lymphatic system disorders) | 3 (3)
muscle cramps (Musculoskeletal and connective tissue disorders) | 8 (8)
musculoskeletal range of motion (Musculoskeletal and connective tissue disorders) | 3 (3)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 4 (4)
nocturia (Renal and urinary disorders) | 2 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 5 (5)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
tremors (General disorders) | 2 (2)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 3 (3)
weakness (General disorders) | 3 (3)
weight gain (Investigations) | 3 (3)
weight loss (Investigations) | 2 (2)
infection (Infections and infestations) | 3 (3)
UTI (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No